CLINICAL TRIAL: NCT00609947
Title: A Clinical Evaluation of the Medtronic Endeavor Zotarolimus-Eluting Coronary Stent System in the Treatment of De Novo Lesions in Small Diameter Native Coronary Arteries
Brief Title: Endeavor Zotarolimus - Eluting Stent in the Treatment Lesions in Small Native Coronary Arteries.
Acronym: ENDEAVORSVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP057
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endeavor Zotarolimus-Eluting Coronary Stent (Experimental): Zotarolimus-eluting stent (ZES) implanted using standard percutaneous coronary intervention (PCI) technique via the femoral approach
  Interventions: Device: Endeavor Zotarolimus-Eluting Coronary Stent

INTERVENTIONS:
Device: Endeavor Zotarolimus-Eluting Coronary Stent
  Other Names: Endeavor

SUMMARY:
The objective of this study is to verify the safety and efficacy of the Endeavor Zotarolimus-Eluting Coronary Stent System for improving coronary luminal diameter in patients with ischemic heart disease due to de novo lesions of length ≤27 mm in native coronary arteries with reference vessels ≥ 2.25 mm to ≤ 2.75 mm.

ELIGIBILITY:
GENERAL INCLUSION CRITERIA:

* The patient is ≥18 years of age.
* The patient has clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia, or positive functional study.
* The patient is an acceptable candidate for Percutaneous Transluminal Coronary Angiography (PTCA), stenting, and emergent Coronary Artery Bypass Grafting (CABG) surgery.
* Female patients of childbearing potential must have a negative pregnancy test within 7 days before the procedure.
* The patient or patient's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board of the respective clinical site.
* The patient agrees to return to same research facility for all required post-procedure follow-up visits.

ANGIOGRAPHIC INCLUSION CRITERIA

1. The target lesion/vessel must meet the following criteria:

1. The patient requires treatment of either:

   * A single de novo lesion located in a native coronary artery amenable to treatment with a 2.25mm, 2.5mm or 2.75mm stent, or
   * Two de novo lesions located in separate target vessels, with at least one of the target lesions amenable to treatment with a 2.25mm, 2.5mm, or 2.75mm stent and the second lesion amenable to treatment with a 2.25mm, 2.5mm, or 2.75mm stent or a 3.0mm or 3.5mm approved Endeavor stent.
2. The lesion(s) must be ≤ 27mm in length.
3. The lesion(s) must have a stenosis of ≥ 50% and < 100%.
4. The vessel(s) has (have) a thrombolysis in myocardial infarction (TIMI) flow 2 or greater.
5. The target vessel reference diameter must be ≥ 2.25mm and ≤ 2.75mm and the second target vessel reference diameter, if present, must be ≥ 2.25mm and ≤ 3.5mm.
6. All target lesions can be treated with a Medtronic Endeavor stent.

GENERAL EXCLUSION CRITERIA:

1. Known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, ticlopidine, clopidogrel, cobalt, nickel, chromium, molybdenum, polymer coatings, or sensitivity to contrast media, which cannot be adequately pre-medicated
2. History of allergic reaction or significant sensitivity to drugs such as zotarolimus, rapamycin, tacrolimus, everolimus, or any other analogue or derivative
3. Platelet count <100,000 cells/mm³ or >700,000 cells/mm³, or white blood cell count <3,000 cells/mm³
4. Serum creatinine level >2.0 mg/dl within 7 days prior to index procedure
5. Evidence of acute MI within 72 hours of intended index procedure
6. Planned PCI of any vessel within 30 days pre or post-index procedure and/or planned PCI of the target vessel(s) within 12 months post-procedure.
7. During the index procedure, the target lesion(s) requires treatment with a device other than PTCA prior to stent placement
8. History of stroke or transient ischemic attack (TIA) within prior 6 months
9. Active peptic ulcer or upper gastrointestinal (GI) bleeding within prior 6 months.
10. History of bleeding diathesis or coagulopathy or patient will refuse blood transfusions.
11. Concurrent medical condition with life expectancy of less than 12 months.
12. Any previous or planned treatment of target vessel with anti-restenotic therapies including but not limited to brachytherapy.
13. Currently participating in an investigational drug or another device study that has not completed primary endpoint or that clinically interferes with current study endpoints; or requires coronary angiography, IVUS or other coronary artery imaging procedures.
14. Documented left ventricular ejection fraction (LVEF) <30% at most recent evaluation.
15. Inability to comply with protocol required medication regimen ANGIOGRAPHIC EXCLUSION CRITERIA

1. Target lesion(s) located in native vessel distal to anastomosis with saphenous vein graft or a left/right internal mammary artery bypass with >40% diameter stenosis anywhere within graft.

2. Previous stenting in the target vessel(s) unless the following conditions are met:

a. It has been at least 9 months since the previous stenting, and b. The target lesion(s) is/are at least 15mm away from the previously placed stent.

3. Target vessel has other lesions with >40% diameter stenosis based on visual estimate or on-line QCA 4. Target vessel(s) has/have evidence of thrombus 5. Target vessel(s) is excessively tortuous (two bends ≥90º to reach target lesion) 6. Target lesion has any of the following characteristics:

1. Location is aorto-ostial, an unprotected left main lesion, or within 5 mm of the origin of the left anterior descending (LAD), left circumflex (LCX), or right coronary artery (RCA)
2. Involves a side branch >2.0 mm in diameter
3. Is at or distal to a >45º bend in the vessel
4. Is severely calcified
5. Involves a bifurcation 7. Unprotected left main coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2008-01; Primary Completion 2012-03 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, Principal Investigator — Columbia University
Locations (1):
- AnMed Health Medical Center, Anderson, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by local and regional medical centers from December 21, 2007 through November 22, 2010.
Pre-assignment Details: Subjects were excluded from participation if they did not meet inclusion/exclusion criteria and fall into the category of per protocol small vessel stenting - 2.25mm, 2.5mm and 2.75mm - single or multi-vessel (Rev K).
Groups:
- Endeavor Zotarolimus-Eluting Coronary Stent: Zotarolimus-eltuing stent (ZES) implanted using standard percutaneous coronary intervention (PCI) technique via the femoral approach
Period: Overall Study
Arm/Group | Endeavor Zotarolimus-Eluting Coronary Stent
Started | 241
Completed | 240 (One death due to automobile accident.)
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Endeavor Zotarolimus-Eluting Coronary Stent
Number analyzed (Participants) | 241
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 231
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 156
Region of Enrollment [Number; unit: participants]
  United States | 241

OUTCOME MEASURES:

1. Primary Outcome: In-segment Percent Diameter Stenosis at 8 Months Post-procedure
Description: In-segment percent diameter stenosis at 8 months post-procedure with percent diameter stenosis defined as the value calculated as 100 x (RVD - Minimal Lumen Diameter (MLD)/RVD using the mean values from two orthogonal views (when possible) by Qualitative Coronary Angiography (QCA).
Time Frame: 8 months post-procedure
Population: The primary analysis sample consisted of 176 subjects (ITT) including the first 97 subjects with 2.25 mm, 39 subjects with 2.50 mm and 40 subjects with 2.75mm stents who met the study entry criteria, signed the written informed consent, and were enrolled in the trial.
Measure: Mean (95% Confidence Interval); unit: percent diameter stenosis
Groups:
- Primary Effectiveness Analysis Endpoint - SVS: The 8-month in-segment diameter stenosis from Endeavor Small Vessel Study (SVS) subects
Arm/Group | Primary Effectiveness Analysis Endpoint - SVS
Number analyzed (Participants) | 176
percent diameter stenosis | 37.4 [16.6 to 58.2]
Statistical Analysis 1: Comparison: Primary Effectiveness Analysis Endpoint - SVS; The 8-month in-segment percent diameter stenosis from Endeavor SVS subjects was compared to the 6-month in-segment percent diameter stenosis from Micro Driver subjects. This study assessed the superiority of SVS against the Micro-Driver regarding in-segment percent diameter stenosis at 8 months post procedure; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The null and alternative hypotheses were: H0: µSVS ≥µM H1: µSVS < µM where µSVS was the mean in-segment 8-month percent diameter stenosis for the SVS study and µM was the mean in-segment 6-month percent diameter stenosis for Micro-Driver; The sample size was not reduced below 158 evaluable subjects in order to support the analysis of the primary safety endpoint; Mean Difference (Final Values) = 49.2, Standard Deviation 21.8

2. Primary Outcome: Major Adverse Cardiac Events (MACE) Rate
Description: Major Adverse Cardiac Events rate at 12 months post-procedure defined as death, target-vessel Myocardial Infarction (Q wave and non-Q wave), emergent cardiac bypass surgery, or target lesion revascularization, repeat percutaneous transluminal coronary angioplasty or cardiac bypass surgery.
Time Frame: 12 months post-procedure
Population: 12-month MACE Rate was compared to a 20% performance goal.
  * 1st 97 subjects enrolled and implanted with 2.25mm stents
  * 1st 39 subjects enrolled and implanted with 2.5mm stents
  * 1st 40 subjects enrolled and implanted with 2.75mm stents
  * A supplemental safety analysis group of subjects with 2.25mm stents N=38 (included in 2.25mm group N=135)
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Primary Analysis Endpoint
Number analyzed (Participants) | 241
Percentage | 10.0 [10.0 to 13.8]
Statistical Analysis 1: Comparison: Primary Analysis Endpoint; The null and alternative hypotheses of interest are: H0: xSVS >= 20% vs. H1: xSVS < 20%, where x is the true SVS 12-month MACE rate. The assessment of the null hypothesis will be carried out at the one-sided 0.05 level of significance. Rejection of the null hypothesis indicates the SVS 12-month MACE rate is significantly below 20%; Test type: Superiority or Other; p = 0.0041, t-test, 1 sided; Cox Proportional Hazard = 13.5, 95% CI 1-sided [upper limit 20], Standard Error of Mean 6.5

ADVERSE EVENTS:
Time Frame: 1 Year
Groups:
- Primary Analysis Endpoint: * The first 97 subjects enrolled and implanted with 2.25mm stents
  * The first 39 subjects enrolled and implanted with 2.5mm stents
  * The first 40 subjects enrolled and implanted with 2.75mm stents
  * A supplemental safety analysis group of subjects with 2.25mm stents N=38 (included in 2.25mm group N=135)
Arm/Group | Primary Analysis Endpoint
Serious Adverse Events (participants affected / at risk) | 87/176
Other Adverse Events (participants affected / at risk) | 0/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Analysis Endpoint (N=176)
Anaemia (Blood and lymphatic system disorders) | 2 (87)
Accute myocardial infarction (Cardiac disorders) | 3 (87)
angina pectoris (Cardiac disorders) | 10 (87)
angina unstable (Cardiac disorders) | 4 (87)
Atrial Fibrillation (Cardiac disorders) | 3 (87)
Bradycardia (Cardiac disorders) | 1 (87)
Cardiac failure congestive (Cardiac disorders) | 1 (87)
Coronary artery disease (Cardiac disorders) | 6 (87)
Coronary artery dissection (Cardiac disorders) | 1 (87)
Coronary artery occlusion (Cardiac disorders) | 4 (87)
Cronary artery restenosis (Cardiac disorders) | 2 (87)
Coronary artery stenosis (Cardiac disorders) | 11 (87)
In-stent coronary artery restenosis (Cardiac disorders) | 16 (87)
Myocardial infarction (Cardiac disorders) | 1 (87)
Ventricular tachycardia (Cardiac disorders) | 1 (87)
Abdominal pain (Gastrointestinal disorders) | 1 (87)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (87)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (87)
Obstruction gastric (Gastrointestinal disorders) | 1 (87)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1 (87)
Vomiting (Gastrointestinal disorders) | 1 (87)
chest discomfort (General disorders) | 1 (87)
Chest pain (General disorders) | 16 (87)
Injection site haematoma (General disorders) | 1 (87)
Non-cardiac chest pain (General disorders) | 4 (87)
Cholelithiasis (Hepatobiliary disorders) | 1 (87)
Cellulitis (Infections and infestations) | 2 (87)
Infected skin ulcer (Infections and infestations) | 1 (87)
Infection (Infections and infestations) | 1 (87)
Pneumonia (Infections and infestations) | 5 (87)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (87)
injury (Injury, poisoning and procedural complications) | 1 (87)
Pocket erosion (Injury, poisoning and procedural complications) | 1 (87)
Blood creatinine increased (Investigations) | 1 (87)
diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (87)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (87)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (87)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (87)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (87)
Cerebrovascular accident (Nervous system disorders) | 2 (87)
Syncope (Nervous system disorders) | 3 (87)
Transient ischaemic attack (Nervous system disorders) | 1 (87)
Depression (Psychiatric disorders) | 1 (87)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (87)
Renal failure (Renal and urinary disorders) | 1 (87)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (87)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (87)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (87)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (87)
Coronary revascularisation (Surgical and medical procedures) | 1 (87)
Embolism (Vascular disorders) | 1 (87)
Hypertension (Vascular disorders) | 1 (87)
Hypotension (Vascular disorders) | 2 (87)
Intermittent claudication (Vascular disorders) | 1 (87)
Lymphoedema (Vascular disorders) | 1 (87)
Peripheral ischaemia (Vascular disorders) | 1 (87)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No